CLINICAL TRIAL: NCT02460549
Title: Feasibility Study of an Intervention Therapeutic Education for Patients Treated With Androgen Deprivation
Acronym: Nutriprophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-04; 2013-A01169-36 (Other: Agence Nationale de Sécurité du Médicament)
Record Dates: First submitted 2014-04-15; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
Keywords: therapeutic patient education; insulinoresistance; empowerment; prostate cancer; oral endocrine therapy; side effects
MeSH Terms: conditions — Prostatic Neoplasms; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- therapeutic education program (Experimental): patients attend three sessions of therapeutic education
  Interventions: Behavioral: therapeutic education program

INTERVENTIONS:
Behavioral: therapeutic education program

SUMMARY:
The purpose of the study is to build and assess the feasibility of a therapeutic education program, constructed in collaboration with the urologists of the University Hospital of Saint Etienne. The aim of this therapeutic education program is to delay the onset or to reduce the amplitude of the development of insulin resistance and side effects of androgen deprivation therapy in patients treated with androgen deprivation in the context of an evolutive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients supported in consultation Urology at the University Hospital North Saint Etienne.
* Aged over 18 years
* Having an evolutive prostate cancer
* Patient treated with LHRH agonist for at least 6 months - Affiliated with the national health insurance system
* And having completed the worksheet informed consent to participate in the program.

Exclusion Criteria:

* Refusal of participation, protected or under guardianship patients.
* Patients unable to understand the study or unable to follow the educational sessions.
* Patient (s) with documented cognitive or psychiatric history.
* Geographical remotness (more than 100 Kms.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who refused to participate | 6 months

SECONDARY OUTCOMES:
Number of patients in all sessions | 6 months
Number of withdrawals | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne Terrier, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CHU Saint-Etienne, Saint-Etienne
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

REFERENCES:
- [Background] Bolla M, de Reijke TM, Van Tienhoven G, Van den Bergh AC, Oddens J, Poortmans PM, Gez E, Kil P, Akdas A, Soete G, Kariakine O, van der Steen-Banasik EM, Musat E, Pierart M, Mauer ME, Collette L; EORTC Radiation Oncology Group and Genito-Urinary Tract Cancer Group. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med. 2009 Jun 11;360(24):2516-27. doi: 10.1056/NEJMoa0810095. PMID 19516032
- [Background] Golant M, Altman T, Martin C. Managing cancer side effects to improve quality of life: a cancer psychoeducation program. Cancer Nurs. 2003 Feb;26(1):37-44; quiz 45-6. doi: 10.1097/00002820-200302000-00005. PMID 12556711
- [Background] Diefenbach MA, Butz BP. A multimedia interactive education system for prostate cancer patients: development and preliminary evaluation. J Med Internet Res. 2004 Jan 21;6(1):e3. doi: 10.2196/jmir.6.1.e3. PMID 15111269
- [Background] Perol D, Toutenu P, Lefranc A, Regnier V, Chvetzoff G, Saltel P, Chauvin F. [Therapeutic education in oncology: involving patient in the management of cancer]. Bull Cancer. 2007 Mar;94(3):267-74. French. PMID 17371769
- [Background] Rebillard X, Grosclaude P, Lebret T, Patard JJ, Pfister C, Richaud P, Rigaud J, Salomon L, Soulie M. [Projected incidence and mortality from urologic cancer in France in 2010.]. Prog Urol. 2010 Nov;20 Suppl 4:S211-4. doi: 10.1016/S1166-7087(10)70041-5. No abstract available. French. PMID 21129643
- [Background] Crook JM, O'Callaghan CJ, Duncan G, Dearnaley DP, Higano CS, Horwitz EM, Frymire E, Malone S, Chin J, Nabid A, Warde P, Corbett T, Angyalfi S, Goldenberg SL, Gospodarowicz MK, Saad F, Logue JP, Hall E, Schellhammer PF, Ding K, Klotz L. Intermittent androgen suppression for rising PSA level after radiotherapy. N Engl J Med. 2012 Sep 6;367(10):895-903. doi: 10.1056/NEJMoa1201546. PMID 22931259
- [Background] Alibhai SM, Gogov S, Allibhai Z. Long-term side effects of androgen deprivation therapy in men with non-metastatic prostate cancer: a systematic literature review. Crit Rev Oncol Hematol. 2006 Dec;60(3):201-15. doi: 10.1016/j.critrevonc.2006.06.006. Epub 2006 Jul 24. PMID 16860998
- [Background] Hoffmann P, Schulman C. Complications of androgen-deprivation therapy in prostate cancer: the other side of the coin. BJU Int. 2009 Apr;103(8):1020-3. doi: 10.1111/j.1464-410x.2008.08293.x. No abstract available. PMID 19348058
- [Background] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748
- [Background] Shahinian VB, Kuo YF, Freeman JL, Goodwin JS. Risk of fracture after androgen deprivation for prostate cancer. N Engl J Med. 2005 Jan 13;352(2):154-64. doi: 10.1056/NEJMoa041943. PMID 15647578
- [Background] Herr HW, O'Sullivan M. Quality of life of asymptomatic men with nonmetastatic prostate cancer on androgen deprivation therapy. J Urol. 2000 Jun;163(6):1743-6. PMID 10799173
- [Background] Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol. 2006 Sep 20;24(27):4448-56. doi: 10.1200/JCO.2006.06.2497. PMID 16983113
- [Background] Saigal CS, Gore JL, Krupski TL, Hanley J, Schonlau M, Litwin MS; Urologic Diseases in America Project. Androgen deprivation therapy increases cardiovascular morbidity in men with prostate cancer. Cancer. 2007 Oct 1;110(7):1493-500. doi: 10.1002/cncr.22933. PMID 17657815
- [Background] Tsai HK, D'Amico AV, Sadetsky N, Chen MH, Carroll PR. Androgen deprivation therapy for localized prostate cancer and the risk of cardiovascular mortality. J Natl Cancer Inst. 2007 Oct 17;99(20):1516-24. doi: 10.1093/jnci/djm168. Epub 2007 Oct 9. PMID 17925537
- [Background] D'Amico AV, Denham JW, Crook J, Chen MH, Goldhaber SZ, Lamb DS, Joseph D, Tai KH, Malone S, Ludgate C, Steigler A, Kantoff PW. Influence of androgen suppression therapy for prostate cancer on the frequency and timing of fatal myocardial infarctions. J Clin Oncol. 2007 Jun 10;25(17):2420-5. doi: 10.1200/JCO.2006.09.3369. PMID 17557956